CLINICAL TRIAL: NCT02788942
Title: The Relationship Between the Removing Port of the Laparoscopic Cholecystectomy Material and the Port Site Infections
Brief Title: The Removing Port of the Laparoscopic Cholecystectomy Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, M.D., Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Trochar
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Wound Infection
Keywords: Port; Infection; cholecystectomy
MeSH Terms: conditions — Wound Infection; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umbilical (No Intervention): The cholecystectomy material will be removed from umbilical port as usual. This will be control group. Port site infection rates will be measured.
- Epigastric (Experimental): The cholecystectomy material will be removed from epigastric port. This will be experimental group. Port site infection rates will be measured.
  Interventions: Procedure: Removing from Epigastric port

INTERVENTIONS:
Procedure: Removing from Epigastric port — The cholecystectomy material will be removed from epigastric port. This will be experimental group. Port site infection rates will be measured
  Arms: Epigastric

SUMMARY:
Laparoscopic cholecystectomy is gold standard for gallstones. In this study the investigators are investigating the effect of the removing of cholecystectomy material from different ports, to the port site infections.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is gold standard for gallstones. But there is no consensus about which port place is optimal for the removing of the cholecystectomy material from the abdomen. There are different port site infections rates in the literature. The minimal tissue damage of laparoscopic cholecystectomy suggests a lower risk of wound infection, but there are series with an infection range of 8 %. The investigators are investigating is there any difference at the port site infection rates when the cholecystectomy material removed from different ports from the abdomen at the laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has cholelithiasis

Exclusion Criteria:

* Subject has perforated gallbladder
* Subject has malignancy
* Subject has increasing wall thickness of the gallbladder
* Subject has malignancy in the preoperative ultrasonography in the gallbladder
* Subject has pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Port site infections | 2 days
  The cholecystectomy material will be removed from umbilical port at the control group, from the epigastric port at the experimental group. The port site infection rates will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Kaya, Principal Investigator — Sisli Etfal Training and Research Hospital
Locations (1):
- Sisli Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Once a three months time

REFERENCES:
- [Result] Comajuncosas J, Hermoso J, Jimeno J, Gris P, Orbeal R, Cruz A, Pares D. Effect of bag extraction to prevent wound infection on umbilical port site wound on elective laparoscopic cholecystectomy: a prospective randomised clinical trial. Surg Endosc. 2017 Jan;31(1):249-254. doi: 10.1007/s00464-016-4965-z. Epub 2016 May 13. PMID 27177957
- [Result] Farooq U, Rashid T, Naheed A, Barkat N, Iqbal M, Sultana Q. COMPLICATIONS OF LAPAROSCOPIC CHOLECYSTECTOMY: AN EXPERIENCE OF 247 CASES. J Ayub Med Coll Abbottabad. 2015 Apr-Jun;27(2):407-10. PMID 26411129
- [Result] Comajuncosas J, Hermoso J, Gris P, Jimeno J, Orbeal R, Vallverdu H, Lopez Negre JL, Urgelles J, Estalella L, Pares D. Risk factors for umbilical trocar site incisional hernia in laparoscopic cholecystectomy: a prospective 3-year follow-up study. Am J Surg. 2014 Jan;207(1):1-6. doi: 10.1016/j.amjsurg.2013.05.010. Epub 2013 Oct 7. PMID 24112669